CLINICAL TRIAL: NCT03035942
Title: Role of Dexamethasone or Ondansetron in the Quality of Recovery After Intrathecal Morphine Administration in Patients Undergoing Lower Limb Surgery.
Brief Title: Quality of Recovery After Dexamethasone, Ondansetron or Placebo Intrathecal Morphine Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Assistant Professor, MD, PhD, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PUCSP 1863886
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-01

CONDITIONS: Fractures, Bone; Nausea and Vomiting, Postoperative; Pruritus; Morphine Adverse Reaction; Satisfaction, Personal
Keywords: Intrathecal morphine; Nausea and vomiting; Quality of recovery; Patient satisfaction; Pruritus; Postoperative pain
MeSH Terms: conditions — Fractures, Bone; Postoperative Nausea and Vomiting; Pruritus; Personal Satisfaction; Nausea; Vomiting; Patient Satisfaction; Pain, Postoperative | interventions — Dexamethasone; Ondansetron; O-antigen, Acinetobacter strain 90; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, double-blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group assignments will be sealed in sequentially numbered opaque envelopes that were opened after patient inclusion in the study. All care providers, researchers, and patients will be blinded to group assignments. Study 5-mL syringes will be prepared by a nurse independent of the study. Normal saline (5 mL total volume), dexamethasone (made up to 5 mL with normal saline), or ondansetron 4 mg (made up to 5 mL with normal saline) will be drawn into each syringe which will be offered to the anesthesia provider after the opaque envelope was opened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D Group (Experimental): Dexamethasone 8 mg
  Interventions: Drug: Dexamethasone
- O group (Experimental): Ondansetron 4 mg
  Interventions: Drug: Ondansetron
- S group (Placebo Comparator): Normal saline (5 mL total volume)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8 mg (made up to 5 mL with normal saline) will be drawn into each syringe which will be offered to the anesthesia provider after the opaque envelope was opened and administered immediately after spinal anesthesia was performed.
  Other Names: D Group
  Arms: D Group
Drug: Ondansetron — Ondansetron 4 mg (made up to 5 mL with normal saline) will be drawn into each syringe which will be offered to the anesthesia provider after the opaque envelope was opened and administered immediately after spinal anesthesia was performed.
  Other Names: O Group
  Arms: O group
Drug: Saline — Normal saline (5 mL total volume) will be drawn into each syringe which will be offered to the anesthesia provider after the opaque envelope was opened and administered immediately after spinal anesthesia was performed.
  Other Names: Placebo Group
  Arms: S group

SUMMARY:
The aim of this study is to evaluate not only the occurrence of side effects, but the quality of the recovery (QoR-40 Questionnaire) of patients submitted to spinal anesthesia with administration of low doses (0.1 mg) of intrathecal morphine for the surgical treatment of fractures in one of the lower limbs and who will receive prophylactic ondansetron (4mg), dexamethasone (8mg) or placebo.

DETAILED DESCRIPTION:
This randomised, double-blinded trial was approved by the Research Ethics Committee of the School of Medical and Health Sciences, Pontifical Catholic University of São Paulo (Sorocaba, São Paulo - Brazil), on June 14 2016, CAAE (Presentation Certificate for Ethical Appreciation) 58208015.7.0000.5373 (Chairperson Prof. J.A. Costa). On the day of surgery, after completion of the pre-anesthetic evaluation and due explanations of the study, consent will be obtained. No participant will take any pre-anesthetic medication before surgery. Subjects will be randomised using a computer-generated (www.random.org) table of random numbers into 3 groups: S (saline), D (dexamethasone 8 mg), or O (ondansetron 4 mg). Group assignments will be sealed in sequentially numbered opaque envelopes that were opened after patient inclusion in the study. All care providers, researchers, and patients will be blinded to group assignments. Study 5-mL syringes will be prepared by a nurse independent of the study. Normal saline (5 mL total volume), dexamethasone (made up to 5 mL with normal saline), or ondansetron 4 mg (made up to 5 mL with normal saline) will be drawn into each syringe which will be offered to the anesthesia provider after the opaque envelope was opened.

After arrival in the operating room, standard ASA (American Society of Anesthesiologists) monitors will be applied. Immediately after venoclysis,e.v. midazolam will be administered as titrated doses to achieve 3 or 4 on Ramsay scale. Spinal puncture will be performed with the patient in the seated position in the median or paramedian line at L3-L4 or L2-L3 interspace using a 26-gauge Quincke needle. Anesthesia will be established with a single bolus of 0.5% hyperbaric bupivacaine (17.5 mg if ≥ 70 kg or expected surgery duration > 150 minutes and 15 mg if < 70 kg) and preservative-free morphine 0.1 mg. Normal saline will be used for fluid replacement therapy. In case of failure of spinal anesthesia, the technique will be repeated or a general approach will be performed and the patient will be excluded from the study. Titrated doses of midazolam (up to 10 mg) or propofol continuous infusion will be administered to achieve perioperative sedation (≥4 on Ramsay scale). Supplemental oxygen 5 L/min via a vent mask will be administered during and after surgery.

Postanesthesia care unit (PACU) All patients will be transferred to the PACU. Data related to the occurrence of pain, nausea, vomiting, pruritus, urinary retention and time to Aldrete score ≥ 9 at the PACU will be recorded. Pain will be assessed every 15 minutes using a 0-10 numeric pain rating scale (NRS), where zero meant no pain and 10 the worst imaginable pain. Morphine (1 to 2 mg) was administered intravenously every 10 minutes to maintain the pain score below 4 (1 mg when the pain score was <7 and 2 mg when it was ≥7). Postoperative nausea and vomiting (PONV) will be treated with dimenhydrinate (30 mg) intravenously. Pruritus will be classified as follow: 0 - no symptoms, 1 - 3 - mild symptoms, 3 - 7 moderate symptoms and 7 - 10 - severe symptoms. Nalbuphine 5 mg intravenously will be administered when score > 4.

Ward Following discharge from the PACU (minimum stay 60 minutes and Aldrete score ≥ 9), all of the participants were given ketoprofen (100 mg) every 12 hours and dipyrone (30 mg.kg-1, maximum 1 g) every six hours intravenously. Whenever patients judged that their analgesia was insufficient, tramadol (100 mg) was administered intravenously at eight-hour minimum intervals as needed. Postoperative nausea and vomiting (PONV) were treated with dimenhydrinate (30 mg) intravenously. An investigator who was blinded to group assignment collected all postoperative outcome data 24 hours after surgical procedure. Subjects were asked to rate the higher score of pain (NRS) during the hospital ward stay. Tramadol consumption, occurrence of urinary retention and the number of nausea and vomiting episodes were also recorded. These findings were confirmed with the ward nursing staff. All subjects stayed at hospital for at least 24 hours.

Data Collection The baseline QoR-40 questionnaire was completed by the subjects after informed consent was obtained in the preoperative holding area and 24 hours after surgery by a blinded investigator. The QoR-40 questionnaire evaluates five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item was rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-40 ranges from 40 (very poor quality of recovery) to 200 (best quality of recovery).

The primary outcome of interest will be the QoR-40 score on postoperative day 1 (POD1).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II, who will scheduled to undergo surgical treatment of lower limb fractures

Exclusion Criteria:

Patients who:

(i) refused to participate in the study;

(ii) were not able to communicate due to alterations in the level of consciousness, or neurologic, or psychiatric disease;

(iii) presented with contraindication to any of the drugs used in the present study;

(iv) had history of alcohol or drug abuse and

(v) had surgery in the last 10 days were excluded.

Reasons for exclusion after randomisation will be protocol violations or if the anesthesia technique was changed from a spinal to a general approach.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo T Moro, Professor, Principal Investigator — PUC São Paulo University
Locations (1):
- Santa Lucinda Hospital, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobson L, Chabal C, Brody MC, Ward RJ, Wasse L. Intrathecal methadone: a dose-response study and comparison with intrathecal morphine 0.5 mg. Pain. 1990 Nov;43(2):141-148. doi: 10.1016/0304-3959(90)91066-R. PMID 2087326
- [Background] Slappendel R, Weber EW, Dirksen R, Gielen MJ, van Limbeek J. Optimization of the dose of intrathecal morphine in total hip surgery: a dose-finding study. Anesth Analg. 1999 Apr;88(4):822-6. doi: 10.1097/00000539-199904000-00026. PMID 10195531
- [Background] Koju RB, Gurung BS, Dongol Y. Prophylactic administration of ondansetron in prevention of intrathecal morphine-induced pruritus and post-operative nausea and vomiting in patients undergoing caesarean section. BMC Anesthesiol. 2015 Feb 17;15:18. doi: 10.1186/1471-2253-15-18. PMID 25971957
- [Background] Braga AA, Frias JA, Braga FS, Poterio GB, Hirata ES, Torres NA. Spinal anesthesia for cesarean section. Use of hyperbaric bupivacaine (10mg) combined with different adjuvants. Rev Bras Anestesiol. 2012 Nov-Dec;62(6):775-87. doi: 10.1016/S0034-7094(12)70178-2. PMID 23176986
- [Background] Krajnik M, Zylicz Z. Understanding pruritus in systemic disease. J Pain Symptom Manage. 2001 Feb;21(2):151-68. doi: 10.1016/s0885-3924(00)00256-6. PMID 11226766
- [Background] Griffiths JD, Gyte GM, Paranjothy S, Brown HC, Broughton HK, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007579. doi: 10.1002/14651858.CD007579.pub2. PMID 22972112
- [Background] Wu JI, Lo Y, Chia YY, Liu K, Fong WP, Yang LC, Tan PH. Prevention of postoperative nausea and vomiting after intrathecal morphine for Cesarean section: a randomized comparison of dexamethasone, droperidol, and a combination. Int J Obstet Anesth. 2007 Apr;16(2):122-7. doi: 10.1016/j.ijoa.2006.11.004. Epub 2007 Feb 1. PMID 17275282
- [Background] Szarvas S, Chellapuri RS, Harmon DC, Owens J, Murphy D, Shorten GD. A comparison of dexamethasone, ondansetron, and dexamethasone plus ondansetron as prophylactic antiemetic and antipruritic therapy in patients receiving intrathecal morphine for major orthopedic surgery. Anesth Analg. 2003 Jul;97(1):259-63, table of contents. doi: 10.1213/01.ane.0000066310.49139.2a. PMID 12818978
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | O Group | D Group | S Group
Started | 45 | 45 | 45
Completed | 37 | 41 | 40
Not Completed | 8 | 4 | 5
Not completed — Adverse Event | 8 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | O Group | D Group | S Group | Total
Number analyzed (Participants) | 37 | 41 | 40 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 41 | 40 | 118
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [24 to 47] | 40 [26 to 54] | 35 [25 to 49] | 40 [25 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 11 | 35
  Male | 24 | 30 | 29 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 37 | 41 | 40 | 118
ASA status [Count of Participants; unit: Participants]
  Physical status ASA 1 (health person) | 23 | 21 | 11 | 55
  Physical status ASA 2 (mild systemic disease) | 14 | 20 | 29 | 63
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 25 [24 to 28] | 26 [24 to 28] | 27 [24 to 29] | 26 [24 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery
Description: Quality of Recovery Questionnaire (QoR-40). Minimum score 40 (very poor quality of recovery) and maximun score 200 (excellent quality of recovery). Higher scores mean better outcome
Time Frame: Twenty four hours after surgery by a blinded investigator
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | O Group | D Group | S Group
Number analyzed (Participants) | 37 | 41 | 40
Score on a scale | 184 [179 to 195] | 187 [181 to 196] | 185 [176 to 196]

2. Secondary Outcome: Nausea and Vomiting During PACU Staying
Description: The occurrence of PONV will be registered during the PACU
Time Frame: 4h
Measure: Count of Participants; unit: Participants
Arm/Group | O Group | D Group | S Group
Number analyzed (Participants) | 37 | 41 | 40
Participants | 3 | 9 | 9

3. Secondary Outcome: Number of Participants With Pruritus
Description: The occurrence of localized or generalized itching (patients who answered yes or no)
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | O Group | D Group | S Group
Number analyzed (Participants) | 37 | 41 | 40
Participants | 4 | 7 | 8

4. Secondary Outcome: Pain During Postanesthesia Care Unit and Ward Stay (Numeric Rating Scale - NRS)
Description: Pain were assessed every 15 minutes during postanesthesia care unit, where zero meant no pain and 10 the worst imaginable pain (higher values represent worse outcome). Twenty four hours after surgery, patients were asked to describe the highest pain score (NRS) during ward stay.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Score on a scale (NRS)
Arm/Group | D Group | O Group | S Group
Number analyzed (Participants) | 37 | 41 | 40
Score on a scale (NRS) | 0 [0 to 5] | 5 [3 to 7] | 2 [0 to 6]

ADVERSE EVENTS:
Time Frame: One week
Description: The occurrence of fail of spinal anesthesia, allergic reactions, urinary retention, respiratory depression were recorded.
Arm/Group | D Group | O Group | S Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 4/45 | 8/45 | 5/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D Group (N=45) | O Group (N=45) | S Group (N=45)
Fail of spinal anesthesia (Surgical and medical procedures) | 4 (4) | 8 (8) | 5 (5) — A second attempt was necessary or the technique was changed to general anesthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03035942/SAP_001.pdf
  • Study Protocol (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03035942/Prot_002.pdf